CLINICAL TRIAL: NCT02992405
Title: Evaluation of Feasibility and Effect Size of a Resilience Enhancement Program for Couples and Families Contending With Cancer (FOCUS)
Brief Title: FOCUS:Families OverComing Under Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, William Saltzman, Psychologist, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT2016-02-SALTZMAN-FOCUS
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Cancer; Depression; PostTraumatic Stress Disorder; Anxiety
MeSH Terms: conditions — Neoplasms; Depression; Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — Therapeutics; Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOCUS Resilience Enhancement Program (Experimental): Those assigned to the immediate treatment group will participate in the 10-week treatment.
  Interventions: Behavioral: FOCUS Resilience Enhancement Program
- Waitlist Treatment (Experimental): After the 10-week immediate treatment period, wait-list control participants will be administered the treatment.
  Interventions: Behavioral: Waitlist (No Study Treatment)

INTERVENTIONS:
Behavioral: FOCUS Resilience Enhancement Program — Each couple or family will have 10 weekly 75 minute sessions comprising the treatment protocol.Questionnaires will be administered at baseline-before the immediate treatment phase (T1) and after the 10-week treatment is completed (T2).
  Other Names: Therapy
  Arms: FOCUS Resilience Enhancement Program
Behavioral: Waitlist (No Study Treatment) — Participants assigned to the Waitlist (No Treatment) group will receive the study intervention only after the 10 weeks of the immediate treatment phase has been completed. Questionnaires will be administered at baseline-before the immediate treatment phase (T1) and after the immediate treatment phase is completed (T2).
  Arms: Waitlist Treatment

SUMMARY:
The FOCUS program (study treatment) is an established evidence-based intervention whose redesign for families and couples dealing with serious and chronic illnesses will provide a creative and promising supplement to the existing support services at Cedars-Sinai Medical Center. All participants will receive the 10-weeks of 75-minute weekly study treatment, but will be split into two groups, the immediate treatment group and the wait list treatment group, who will receive the study treatment after the immediate 10 weeks of treatment is completed.

DETAILED DESCRIPTION:
Despite advances in the development of brief evidence-based programs for families and couples contending with illness, trauma or loss, the support services provided at even top-tier medical facilities are overwhelmingly focused on the individual patient. In most cases, combined treatment with spouses and family members is the exception rather than the rule.

FOCUS is one of the very few programs that has a strong evidence base and has been used in medical settings. It is a preventive, skill-based training program that is customized for each couple or family and is designed to build upon existing strengths in order to enhance family and individual resilience.

A cancer diagnosis is a family affair. Research has shown that the family or spousal relationship can be instrumental in lessening patient distress and supporting treatment compliance and positive adjustment across the various stages of treatment, survivorship, recurrence / relapse, and end-of-life. Reductions in patient depression and anxiety through couple or family interventions may reduce overall healthcare utilization and cost while improving care quality.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent will be obtained from each participating adult subject and written assent from each minor participating in the program. Specific criteria for inclusion into the program are as follows:

1. Couples must have at least one partner and families at least one parent who is or has been diagnosed with cancer at least 30 days prior to study start and not more than one year from last treatment visit.
2. Couples or parents must be at least 18 years old and must be English speakers.
3. At least one member of the couple must score >60 on the Anxiety or Depression scale on the Brief Symptom Index 18 administered during the screening visit and/or have notable difficulties in relationship or family functioning, as resulted in a ≥2 score in FAD subscale or at least one RDAS subscale question answered 'more often than not' or more frequent.
4. The families participating in the study must have at least one child older than the age of five.
5. Participating families must have at least one parent who can provide legal consent for the participation of their child(ren) in the program.
6. Participants must be willing and able to complete 10 sessions within 14 weeks.
7. Participants undergoing active management or care plans for abuse or psychopathology may enroll in study if reports of ongoing management are provided.

Exclusion Criteria:

1. There must not be any participant with urgent and/or immediate health needs (where a possible 10-week wait time poses more than minimal risks).
2. There must not be active (within the last 30 days and/or during study intervention) and unmanaged domestic violence or abuse, substance abuse, or extreme forms of psychopathology such as psychosis that would interfere with the treatment.
3. Primary presenting personal and/or relational issues are largely unrelated to the cancer diagnosis and treatment, as determined by the screening clinician.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of program as defined by dropout rate | 10 weeks
  A randomized controlled trial will be considered feasible if the dropout rate is less than or equal to 20%.

SECONDARY OUTCOMES:
Change in score of depression as measured by the Patient Health Questionnaire 9 (PHQ-9). | 10 weeks
Change in score of anxiety as measured by the General Anxiety Disorder 7 (GAD-7). | 10 weeks
Change in score of post traumatic stress as measured by the PTSD Checklist - Civilian (PCL-C). | 10 weeks
Change in score of stress in Human Functioning as measured by the Sense of Coherency (SOC). | 10 weeks
Change in score of quality of life as measured by the Functional Assessment of Cancer Therapy - General Version (FACT-G). | 10 weeks
Change in score of caregiver's quality of life as measured by the Caregiver Quality of Life Index - Cancer (CQOLC). | 10 weeks
Change in score of family functioning as measured by the McMasters Family Assessment Device (FAD). | 10 weeks
Change in score of couples relational functioning as measured by the Revised Dyadic Adjustment Scale (RDAS). | 10 weeks
Change in parents' score of child functioning as measured by the Strengths and Difficulties Questionnaire (SDQ). | 10 weeks
Change in patient satisfaction score as measured by the FOCUS Impact Rating Scale (FIRS). | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Saltzman, PhD, Principal Investigator — Cedars-Sinal Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States